CLINICAL TRIAL: NCT03471312
Title: Effect of Oral Magnesium Therapy on Constipation on Children With Cerebral Palsy
Brief Title: Effect of Oral Magnesium Therapy on Constipation on Cerebral Palsy Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, NAMostafa, principal investigator, Assiut University
Other Study IDs: constipation on cp patients
Record Dates: First submitted 2018-03-10; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Magnesium Therapy on Cerebral Palsy Patients
MeSH Terms: interventions — Magnesium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- treated with magnesium therapy: will receive magnesium sulphate 10 mg \kg \day as a single oral dose for one month duration
  Interventions: Drug: Magnesium
- treated with placebo drug: will receive placebo drug
  Interventions: Drug: Magnesium

INTERVENTIONS:
Drug: Magnesium — magnesium therapy
  Other Names: placebo

SUMMARY:
The aim of this study is to study the therapeutic and adverse effects of oral magnesium sulfate therapy on constipation in children with spastic cerebral palsy suffering from chronic constipation in neuro pediatric unit at Assiut University Hospital.

DETAILED DESCRIPTION:
Children with cerebral palsy (CP) often experience many comorbidities such as constipation,which is considered a frequent problem in spastic (cp)children .It occurs due to reduced mobility, difficulties in feeding and as a side effect of many muscle relaxing medications.It is estimated that 74% of children with cerebral palsy suffer from constipation ,which necessitates use of laxatives. Magnesium sulfate has a famous role as being an osmotic laxative,which is the first step in the pharmacological treatment of constipation

• Mechanism of action of mg sulphate: They are poorly absorbed by the intestinal wall, which leads to intraluminal accumulation of hyperosmolar particles. This stimulates retention of water in the intestinal lumen, softening the stools and increasing peristalsis through intestinal distension. It acts by accelerating small intestinal transit both in fasting and in fed state and it tends to increase the frequency and weight of stools, compared with placebo.In addition ,It increases intraluminal secretion of cholecystokinin and increases nitric oxide (NO) release.

• Side effects of mg sulphate: Reducing the intestinal absorption of fat, protein and carbohydrates following solid meal ingestion

• other drugs used as laxative in cp and there side effects:

* Lactulose: it can lead to distention, bloating and excess flatus. In some individuals these side-effects may limit the use of this product.
* Glycerin: is another small molecule that can exert osmotic activity in the colon. It is not absorbed by the colon and is used as a suppository to draw water into the rectum to produce a bowel movement. It is well absorbed by the small intestine, and hence cannot be taken by oral route.

  * The aim of this study is to study the therapeutic and adverse effects of oral magnesium sulfate therapy on constipation in children with spastic cerebral palsy suffering from chronic constipation in neuro pediatric unit at Assiut University Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as cerebral palsy
2. Age below18 year
3. Presence of constipation according to ROME criteria

Exclusion Criteria:

1. Patients with cardiac problem
2. Patients with renal problem
3. Patients with GIT problem or chronic diarrhea

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: cerebral palsy patients in the neuro pediatric unit, at Assiut University Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
EVALUATE THE EFFECT OF ORAL MAGNESIUM THERAPY ON CONSTIPATION IN CHILDREN WITH CEREBRAL PALSY BY A QUESTIONNAIRE | baseline
  Evaluate the effect of oral magnesium therapy on constipation in children with spastic cerebral palsy suffering from chronic constipation in neuro pediatric unit at assiut university hospital by comparison of the percentage of improving cases in the 2 groups (first group using oral magnesium therapy . second group using placebo) by a questionnaire asking about amount , frequency and nature of stool

SECONDARY OUTCOMES:
Evaluate the main side effect of oral magnesium therapy (Diarrhea) | baseline
  Evaluate the main side effect of oral magnesium therapy (Diarrhea) on constipation in children with spastic cerebral palsy suffering from chronic constipation in neuro pediatric unit at assiut university hospital by a questionnaire asking about amount , frequency and nature of stool